CLINICAL TRIAL: NCT03074279
Title: Risk Factors in Sudden Unexpected Death in Epilepsy of the Adults and Children: A Matched Case-control Study
Brief Title: Risk Factors of SUDEP
Acronym: PRERIES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: French Foundation for Epilepsy Research (FFRE) (Unknown); The French League Against Epilepsy (LFCE) (Unknown); University Hospital, Bordeaux (Other); University Hospital, Lille (Other); Hospices Civils de Lyon (Other); University Hospital, Marseille (Other); Central Hospital, Nancy, France (Other); Hopital Universitaire Robert-Debre (Other); Rennes University Hospital (Other); University Hospital, Strasbourg, France (Other); ToulouseUniversity Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8601
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; SUDEP; case-control study; risks factors
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patient with epilepsy who died as a result of confirmed or probable SUDEP and NEAR SUDEP during the study period.
  Interventions: Other: Interview with a psychologist and self-reported questionnaires
- Controls: Patient with epilepsy matched by: âge, etiology and type of epilepsy, level of seizure control
  Interventions: Other: Interview with a psychologist and self-reported questionnaires

INTERVENTIONS:
Other: Interview with a psychologist and self-reported questionnaires — The family members or patients who decide to participate in the study will be asked to complete an interview with a psychologist (semistructured interview, standard form, questionnaires) and self-reported questionnaires

SUMMARY:
Numerous studies over the past decade have shown without any doubt that there is a higher mortality risk in patients with epilepsy than in the general population. The cause of death may be related to the cause of epilepsy, being directly related to a seizure (status epilepticus or sudden unexpected death in epilepsy; SUDEP), a consequence of seizures (accidents, etc), other associated pathologies (cancer, cardiovascular disease, ischemic heart disease, pneumonia, etc) or an associated disorder (depression or suicide). A SUDEP is defined as a sudden, non-traumatic, unexpected death in a patient with epilepsy, not necessarily in the presence of witnesses, that is not due to drowning, with or without evidence of a seizure, excluding documented status epilepticus and in which a post-mortem autopsy reveals no anatomical or toxicological cause of death. Little is known about SUDEP and its mechanisms and risk factors.

This epidemiological study is based on the RSME. The Main objective of this study to identify risk factors of SUDEP, in particular night-time supervision and the risks associated with anti-epileptic drugs including compliance and drug interactions.

DETAILED DESCRIPTION:
Numerous studies over the past decade have shown without any doubt that there is a higher mortality risk in patients with epilepsy than in the general population. The cause of death may be related to the cause of epilepsy, being directly related to a seizure (status epilepticus or sudden unexpected death in epilepsy; SUDEP), a consequence of seizures (accidents, etc), other associated pathologies (cancer, cardiovascular disease, ischemic heart disease, pneumonia, etc) or an associated disorder (depression or suicide). A SUDEP is defined as a sudden, non-traumatic, unexpected death in a patient with epilepsy, not necessarily in the presence of witnesses, that is not due to drowning, with or without evidence of a seizure, excluding documented status epilepticus and in which a post-mortem autopsy reveals no anatomical or toxicological cause of death. Little is known about SUDEP and its mechanisms and risk factors.

A French national network on epilepsy related death (Reseau Sentinelle Mortalité Epilepsie, RSME) will be initially established in 2010 by the French League Against Epilepsy (LFCE) under the leadership of bereaved families and supported by the French Foundation for Epilepsy Research (FFRE). This epidemiological study is based on the RSME.

The Main objective of this study to identify risk factors of SUDEP, in particular night-time supervision and the risks associated with anti-epileptic drugs including compliance and drug interactions.

The study design is an epidemiological case-control study. The cases are SUDEP identified in the RSME and French centres of Epileptology.

Epilepsy-related deaths are reported by physicians but also by bereaved families. An interview with a psychologist will be proposed at this moment.

The control group will include patients with epilepsy and relatives of patients from tertiary epilepsy units (in particular, participants of GRENAT registry or a national multicenter study RESPOMSE), private neurologists or general practitioners and thanks from patients associations.

Sociodemographic data, lifestyle, personal and family medical history will be collected during an interview with a psychologist by phone or during a face to face interview. For bereaved families, information on causes and circumstances of beloved one's death will be collected during these interviews.The characteristics of epilepsy will be completed by the patient's neurologist.

ELIGIBILITY:
Inclusion Criteria:

Cases : Any patient with active epilepsy (treated or not) or in remission under treatment or without treatment for at least two years who died as a result of confirmed or probable SUDEP or NEAR SUDEP during the study period.

Controls : Patient with active epilepsy (treated or not) or in remission under treatment or without treatment for at least two years and matched by: age, epileptic syndrom and level of seizure controls

Exclusion Criteria:

For cases and controls :patient not living in France, refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Cases : Confirmed or probable SUDEP or nearSUDEP reported by physicians of the "Réseau Sentinelle Mortalité Epilepsie" (RSME) or by bereaved families. The bereaved families will be contacted by a psychologist who proposes an interview.
  Controls : Patients with epilepsy and relatives of patients recruited from tertiary epilepsy units, private neurologists or general practitioners and thanks from patients associations.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Estimated)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors for SUDEP | 1 day
  * Lifestyle (night-time supervision ...), habits (alcohol consumption ...)
  * Personal cardiac history (arrhythmias, ECG abnormalities ...), respiratory, sleep apnoea, muscular or neurological disorders, mental retardation, associated psychiatric disorders…
  * Antiepileptic drugs

SECONDARY OUTCOMES:
Familial Risk factors for SUDEP | 1 day
  Family history of epilepsy, Family history of sudden death, arrhythmias, sleep apnea
Needs and expectations of bereaved families on epilepsy related death information | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine Picot, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
NC

REFERENCES:
- [Background] Donner EJ, Waddell B, Osland K, Leach JP, Duncan S, Nashef L, Picot MC. After sudden unexpected death in epilepsy: Lessons learned and the road forward. Epilepsia. 2016 Jan;57 Suppl 1:46-53. doi: 10.1111/epi.13235. PMID 26749016